CLINICAL TRIAL: NCT03990883
Title: A Randomized, Subject- and Evaluating Investigator-blinded, Controlled, Multicenter, Split-face, Comparison Clinical Investigation to Evaluate Effectiveness and Safety of Princess FILLER Lidocaine in the Correction of Nasolabial Folds
Brief Title: Effectiveness and Safety of Princess FILLER Lidocaine in Correction of Nasolabial Folds (NLF)
Acronym: FILIDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPH 301-201200F
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-07

CONDITIONS: Dermatological Non-Disease
Keywords: nasolabial folds; correction

STUDY DESIGN:
Intervention Model Description: Pivotal study
Who Masked: Participant, Outcomes Assessor
Masking Description: subject- and evaluator-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment of device 1 on left side (Other): Treatment of nasolabial folds (NLF) with both Investigational Device and Comparator; Princess Filler Lidocaine is assigned to left NLF, Comparator is assigned to right NLF
  Interventions: Device: Princess Filler Lidocaine
- Treatment of device 1 on right side (Other): Treatment of nasolabial folds (NLF) with both Investigational Device and Comparator; Princess Filler Lidocaine is assigned to right NLF, Comparator is assigned to left NLF
  Interventions: Device: Princess Filler Lidocaine

INTERVENTIONS:
Device: Princess Filler Lidocaine — correction of nasolabial folds

SUMMARY:
Clinical Investigation to demonstrate the effectiveness and safety of Princess Filler Lidocaine in the correction of moderate to severe nasolabial folds

DETAILED DESCRIPTION:
Clinical Investigation to assess the effectiveness of "Princess Filler Lidocaine" in reducing the severity of nasolabial folds compared to "Juvederm Ultra XC", based on the independent blinded evaluating investigator live assessment using the Nasolabial Folds Severity Rating Scale (NLF-SRS) at Week 24 after initial treatment and relative to Baseline assessments

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 22 years of age or older, at the Screening visit
2. Subjects with two fully visible, approximately symmetrical moderate to severe NLFs (same severity) with severity scores of 2 or 3 on the 5- point NLF-SRS for both NLF as judged by the treating investigator in conjunction with the independent blinded evaluating investigator.
3. Females of childbearing potential must have a negative urine pregnancy test at injection visits and must agree to use an adequate method of contraception for the duration of the clinical investigation
4. Healthy skin in the nasolabial area and free of diseases that could interfere in cutaneous aging evaluation
5. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of the clinical investigation, including botulinum toxin injections (except glabellar or forehead botulinum toxin treatment)
6. Subjects having understood the purpose and conduct of the clinical investigation and having given written informed consent

Exclusion Criteria:

1. For females: pregnant and/or lactating or planning to become pregnant during the clinical investigation
2. History of allergies or hypersensitivity to HA preparations, lidocaine or anesthetics of any amide-based anesthetic
3. Since Juvéderm® Ultra XC contains trace amounts of Gram-positive bacterial proteins, subjects with history of allergies to such material can not be included in this clinical investigation
4. Tendency to keloid formation, hypertrophic scars and/or pigmentation disorders
5. Known human immune deficiency virus-positive individuals
6. Presence of infectious, inflammatory or proliferative cancerous or pre-cancerous lesions in the area to be treated
7. Re-current herpes simplex in the treatment area
8. History or presence of any autoimmune or connective tissue disease, or current treatment with immunomodulating therapy
9. Uncontrolled (or instable) diabetes mellitus or systemic diseases
10. Facial plastic surgery, tissue augmentation with silicone, fat or another non-absorbable substance (permanent fillers) area of device application
11. Implantation of facial dermal fillers in the treatment area in the preceding twelve months
12. Skin of the nasolabial region affected by aesthetic treatments (e.g. laser therapy, absorbable and non-absorbable sutures (threads), microneedling and/or botulinum toxin within the last twelve months, dermabrasion and mesotherapy within the last six months, chemical peeling within the last three months) or planning to undergo such procedures during the clinical investigation
13. Facial lypolysis, including submental fat treatments, within last month prior to enrollment and during the clinical investigation
14. Bariatric surgery within 12 months prior to enrollement and during the clinical investigation
15. History of bleeding disorders and/or use of anticoagulant, antiplatelet or thrombolytic medication from ten days pre- to three days post injection
16. Planned dental/oral surgery or modification (bridge-work, implants) within two weeks prior injection and to a minimum of four weeks post injection
17. Any medical condition prohibiting the inclusion in the clinical investigation according to the judgment of the treating investigator
18. Previous enrollment in this clinical investigation
19. Current participation in another clinical investigation, or treatment with any investigational drug/medical device within 30 days prior to clinical investigation enrollment
20. Any dependency of the subject to the treating investigator, the blinded independent evaluating investigator or clinical investigation site (e.g. employees of the sponsor), or subjects who are employees or relatives of the treating investigator and/or the independent blinded evaluating investigator
21. Subjects who have one of the following assessments during the visual examinations at Baseline:

Snellen visual acuity test worse than 20/40 (with corrective eyewear, if applicable), abnormal confrontational visual field test, or abnormal ocular motility test.

Repeat Treatment - Inclusion Criteria:

1. In the opinion of the treating investigator, the subject has returned to sufficient severity of both NLFs that would have qualified him for enrollment into the clinical investigation initially (note that the subject does not have to return to his Baseline severity to be permitted to receive a repeat treatment)
2. Subjects with NLFs with severity scores of 2 or 3 on the 5-point NLF-SRS for both NLFs as judged by the treating investigator in conjunction with the independent blinded evaluating investigator (note that it is not necessary for the treating and evaluating investigator to agree on the same rating)
3. Females of childbearing age must have a negative urine pregnancy test at the repeat-treatment visit and must agree to continue to use an adequate method of contraception for the duration of the clinical investigation
4. Healthy skin in the nasolabial area and free of diseases that could interfere in cutaneous aging evaluation and/or injection

Repeat Treatment - Exclusion Criteria:

1. Occurrence of an SAE or adverse event of special interest (AESI; i.e., changes in vision [loss of vision, blurriness, double vision, pain in or around the eye, blindness, blind spots, problems moving the eyes, change in peripheral vision], skin changing color around the eyelids or around the site of injection) during or after the initial injection and/or touch-up injection
2. Subjects who experienced visual changes or other serious medical conditions during or after the initial/touch-up injection
3. Subjects who have one of the following assessments during the visual examinations:

   * Snellen acuity test worse than 20/40 (with corrective eyewear, if applicable)
   * abnormal confrontational visual field test
   * abnormal ocular motility test
4. Subjects who became pregnant since start of the study or are planning to become pregnant during the clinical investigation
5. Known human immune deficiency virus-positive individuals
6. Presence of infectious, inflammatory or proliferative cancerous or pre-cancerous lesions in the area to be treated
7. Development of recurrent herpes simplex in the treatment area since study start
8. Development of any autoimmune or connective tissue disease since start of participation in the study, or current treatment with immunomodulating therapy
9. Development of uncontrolled (or instable) diabetes mellitus or any other systemic disease since study start
10. Development of a bleeding disorder since study start or use of anticoagulant, antiplatelet or thrombolytic medication from ten days pre- to three days post injection
11. Planned dental/oral surgery or modification (bridge-work, implants) within 2 weeks prior to injection and to a minimum of four weeks post injection
12. Any medical condition prohibiting the inclusion for repeat treatment according to the judgement of the treating investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bank, MD, Principal Investigator — Center of Dermatology, Cosmetic and Laser Surgery; Joel Cohen, MD, Principal Investigator — AboutSkin research, LLC; John Joseph, MDE, Principal Investigator — Dr. John Joseph Facial Plastic and Reconstructive Surgery; Gary Monheit, MD, Principal Investigator — Total Skin and Beauty Dermatology Center; Ava Shamban, MD, Principal Investigator — Ava MD; Susan Taylor, MD, Principal Investigator — University of Pennsylvania; Robert Weiss, MD, Principal Investigator — Maryland Laser Skin and Vein; Sabrina Fabi, MD, Principal Investigator — Cosmetic, Lazer, Dermatology; Jeanine Downie, MD, Principal Investigator — Image Dermatology P.C.; Jeremy Green, MD, Principal Investigator — Skin Research Institute; Michael Gold, MD, Principal Investigator — Tennesse Clinical Research Institute
Locations (11):
- United States (11):
  - Gary Monheit, Birmingham, Alabama
  - John Joseph, Beverly Hills, California
  - Sabrina Fabi, San Diego, California
  - Ava Shamban, Santa Monica, California
  - Joel Cohen, Greenwood Village, Colorado
  - Jeremy Green, Coral Gables, Florida
  - Robert Weiss, Hunt Valley, Maryland
  - Jeanine Downie, Montclair, New Jersey
  - The Center for Dermatology Cosmetic and Laser Surgery, New York, New York
  - Susan Taylor, Philadelphia, Pennsylvania
  - Michael Gold, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 295 enrolled participants, 270 met inclusion criteria and were randomized to treatment.
Groups:
- Treatment With Princess Filler Lidocaine on Left Side, Treatment With Comparator on Right Side: Treatment of nasolabial folds (NLF) with both Investigational Device and Comparator.
  Princess Filler Lidocaine: Injection into the nasolabial fold on the left side of the face.
  Comparator: Injection into the nasolabial fold on the right side of the face.
- Treatment With Princess Filler Lidocaine on Right Side, Treatment With Comparator on Left Side: Treatment of nasolabial folds (NLF) with both Investigational Device and Comparator.
  Princess Filler Lidocaine: Injection into the nasolabial fold on the right side of the face.
  Comparator: Injection into the nasolabial fold on the left side of the face.
- Princess Filler Lidocaine Open Label Extension: Princess Filler Lidocaine Open Label Extension where all subjects from Arm 1 and 2 can receive Experimental Treatment to both right and left nasolabial folds.
  Princess Filler Lidocaine: Injection into nasolabial folds on both sides of the face.
Period: Blinded Treatment Phase
Arm/Group | Treatment With Princess Filler Lidocaine on Left Side, Treatment With Comparator on Right Side | Treatment With Princess Filler Lidocaine on Right Side, Treatment With Comparator on Left Side | Princess Filler Lidocaine Open Label Extension
Started | 136 | 134 | 0
Completed | 113 | 111 | 0
Not Completed | 23 | 23 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 7 | 10 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0
Not completed — COVID-19 | 3 | 2 | 0
Not completed — Personal Reasons | 6 | 3 | 0
Not completed — Temporary Hold on Repeat Treatment | 3 | 2 | 0
Period: Open Label Extension Phase
Arm/Group | Treatment With Princess Filler Lidocaine on Left Side, Treatment With Comparator on Right Side | Treatment With Princess Filler Lidocaine on Right Side, Treatment With Comparator on Left Side | Princess Filler Lidocaine Open Label Extension
Started | 0 | 0 | 48 (176 participants who completed the Blinded Treatment Phase did not enroll into the Open Label Extension Phase because they were either not eligible for repeat-treatment while participating in the study or did not want to receive the optional repeat-treatment.)
Completed | 0 | 0 | 46
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Princess Filler Lidocaine on Left Side, Treatment With Comparator on Right Side | Treatment With Princess Filler Lidocaine on Right Side, Treatment With Comparator on Left Side | Total
Number analyzed (Participants) | 136 | 134 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 112 | 219
  >=65 years | 29 | 22 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.65) | 55.0 (9.08) | 55.4 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 131 | 264
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 31 | 60
  Not Hispanic or Latino | 107 | 103 | 210
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 4 | 10
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 14 | 15 | 29
  White | 112 | 114 | 226
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 136 | 134 | 270
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick skin type is a scale that classifies skin based on its reaction to sun exposure, specifically its tendency to burn or tan. It includes six types:
  Type I: very pale white skin, burns without tanning; Type II: white skin, burns and does not tan easily; Type III: fair skin, burns first then tans; Type IV: light brown skin, burns a little and tans easily; Type V: brown skin, easily tans to a darker color and rarely burns; Type VI: dark brown or black skin, never burns but tans darker
  Participants
    Type I | 9 | 3 | 12
    Type II | 36 | 42 | 78
    Type III | 41 | 40 | 81
    Type IV | 32 | 31 | 63
    Type V | 11 | 10 | 21
    Type VI | 7 | 8 | 15
Nasolabial Folds-Severity Rating Scale (NLF-SRS) [Count of Participants; unit: Participants]
  NLF-SRS Left Side of Face: Grade 0 - none/minimal | 0 | 0 | 0
  NLF-SRS Left Side of Face: Grade 1 - mild | 0 | 0 | 0
  NLF-SRS Left Side of Face: Grade 2 - moderate | 56 | 48 | 104
  NLF-SRS Left Side of Face: Grade 3 - severe | 80 | 86 | 166
  NLF-SRS Left Side of Face: Grade 4 - extreme | 0 | 0 | 0
  NLF-SRS Right Side of Face: Grade 0 - none/minimal | 0 | 0 | 0
  NLF-SRS Right Side of Face: Grade 1 - mild | 0 | 0 | 0
  NLF-SRS Right Side of Face: Grade 2 - moderate | 61 | 51 | 112
  NLF-SRS Right Side of Face: Grade 3 - severe | 75 | 83 | 158
  NLF-SRS Right Side of Face: Grade 4 - extreme | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder Status Based on Independent Evaluating Investigator Live Assessment at Week 24 - Full Analysis Dataset
Description: The percentage of responders based on the independent blinded evaluating investigator live assessment at Week 24 after initial treatment and compared to Juvederm® Ultra XC. Responder is defined as having at least one grade improvement over Baseline, on the 5-point Nasolabial Folds-Severity Rating Scale (NLF-SRS). NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
  Hierarchical Testing Procedure:
  This primary outcome measure is assessed first in a hierarchical testing sequence.
Time Frame: Week 24
Population: The population used consists of all randomized subjects who received Princess® FILLER Lidocaine AND the control Juvéderm® Ultra XC at the same visit as initial treatment; if subjects had received only one treatment (only Princess® FILLER Lidocaine or only Juvéderm® Ultra XC) during initial treatment they would have been excluded from the analysis set. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Princess Filler Lidocaine: Treatment with Princess Filler Lidocaine: Injection into the nasolabial fold on either the left or the right side of the face.
- Comparator: Treatment with Comparator: Injection into the nasolabial fold on either the right or the left side of the face.
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 270 | 270
Participants | 222 | 221
Statistical Analysis 1: Comparison: Princess Filler Lidocaine vs Comparator; Test type: Non-Inferiority — The hypothesis to be tested was: H0: pA-pB ≤ d0 versus H1: pA-pB > d0 where, pA is the response rate for Princess® FILLER Lidocaine, pB is the response rate for the Comparator, and d0 is the non-inferiority margin set at -10%. The hypothesis was tested using a 1-sided, McNemar type test at an alpha of 0.025 with a delta of 0.10 (10%). Assuming pA to be 87% and pB to be 88% a sample size of 222 subjects had been calculated to be sufficient to achieve a power of 90%; p < 0.0001, McNemar; Risk Difference (RD) = 0.37, 95% CI 2-sided [-2.96 to 3.7]

2. Primary Outcome: Responder Status Based on Independent Evaluating Investigator Live Assessment at Week 24 - Per Protocol Dataset
Description: The percentage of responders based on the independent blinded evaluating investigator live assessment at Week 24 after initial treatment and compared to Juvederm® Ultra XC. Responder is defined as having at least one grade improvement over Baseline, on the 5-point Nasolabial Folds-Severity Rating Scale (NLF-SRS). NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
  Hierarchical Testing Procedure:
  This is the second outcome measure in the hierarchical testing sequence. Statistical significance for this measure will only be assessed if the first outcome measure achieves statistical significance at the predefined alpha level (0.025).
Time Frame: Week 24
Population: The population used consists of all randomized subjects who received Princess® FILLER Lidocaine AND the control Juvéderm® Ultra XC at the same visit as initial treatment and who had no major protocol deviations. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 224 | 224
Participants | 187 | 187
Statistical Analysis 1: Comparison: Princess Filler Lidocaine vs Comparator; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, McNemar — The threshold for statistical significance is 0.025. A hierarchical approach is used and results are confirmative if all tests previously performed within the hierarchy achieve significance at a one-sided significance level of 0.025; Risk Difference (RD) = 0, 95% CI 2-sided [-3.71 to 3.71]

3. Secondary Outcome: Responder Status Based on Independent Photographic Reviewers Assessment at Week 24 - Full Analysis Dataset
Description: The percentage of responders based on the independent photographic reviewers assessment at Week 24 after initial treatment and compared to Juvederm® Ultra XC and based on photographs. Responder is defined as having at least one grade improvement over Baseline, on the 5-point Nasolabial Folds-Severity Rating Scale (NLF-SRS). NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
  Hierarchical Testing Procedure:
  This is the third outcome measure to be analyzed in the hierarchical testing sequence. Statistical significance for this measure will only be assessed if the first and second outcome measures achieve statistical significance at the predefined alpha level (0.025).
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 270 | 270
Participants | 165 | 173
Statistical Analysis 1: Comparison: Princess Filler Lidocaine vs Comparator; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.025, McNemar — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -2.96, 95% CI 2-sided [-9.99 to 4.07]

4. Secondary Outcome: Responder Status Based on Independent Photographic Reviewers Assessment at Week 24 - Per Protocol Dataset
Description: The percentage of responders based on the independent photographic reviewers assessment at Week 24 after initial treatment and compared to Juvederm® Ultra XC and based on photographs. Responder is defined as having at least one grade improvement over Baseline, on the 5-point Nasolabial Folds-Severity Rating Scale (NLF-SRS). NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
  Hierarchical Testing Procedure:
  This is the fourth outcome measure in the hierarchical testing sequence. Testing for this measure is contingent upon statistical significance being demonstrated for the first three outcome measures at the predefined alpha level (0.025).
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 224 | 224
Participants | 145 | 146
Statistical Analysis 1: Comparison: Princess Filler Lidocaine vs Comparator; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.009, McNemar — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -0.45, 95% CI 2-sided [-8.42 to 7.52]

5. Secondary Outcome: Responder Status Based on Treating Investigator Live Assessment at Week 24 - Full Analysis Set
Description: The percentage of responders based on the treating investigator live assessment at Week 24 after initial treatment and compared to Juvederm® Ultra XC. Responder is defined as having at least one grade improvement over Baseline, on the 5-point Nasolabial Folds-Severity Rating Scale (NLF-SRS). NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
  Hierarchical Testing Procedure:
  This is the fifth outcome measure to be analyzed as part of the hierarchical testing sequence. Statistical significance will be assessed only if the first four outcome measures demonstrate statistical significance at the predefined alpha level (0.025).
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 270 | 270
Participants | 225 | 226
Statistical Analysis 1: Comparison: Princess Filler Lidocaine vs Comparator; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, McNemar — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -0.37, 95% CI 2-sided [-3.85 to 3.11]

6. Secondary Outcome: Responder Status Based on Treating Investigator Live Assessment at Week 24 - Per Protocol Set
Description: The percentage of responders based on the treating investigator live assessment at Week 24 after initial treatment and compared to Juvederm® Ultra XC. Responder is defined as having at least one grade improvement over Baseline, on the 5-point Nasolabial Folds-Severity Rating Scale (NLF-SRS). NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
  Hierarchical Testing Procedure:
  This is the sixth outcome measure to be analyzed as part of the hierarchical testing sequence. Statistical significance will be assessed only if the first five outcome measures demonstrate statistical significance at the predefined alpha level (0.025).
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 224 | 224
Participants | 194 | 195
Statistical Analysis 1: Comparison: Princess Filler Lidocaine vs Comparator; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, McNemar — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -0.45, 95% CI 2-sided [-4.05 to 3.16]

7. Secondary Outcome: Improvement Over Baseline Based on Independent Blinded Evaluating Investigator Assessment at Week 24
Description: The percentage of subjects with an improvement over Baseline (subjects who have been rated as "very much improved" or "much improved" or "improved"), based on the independent blinded evaluating investigator assessment at Week 24 after initial treatment and using the 5-point Global Aesthetic Improvement Scale (GAIS). GAIS grades are ranked as "very much improved", "much improved", "improved", "no change", and "worse".
Time Frame: Week 24
Population: The population used consists of all randomized subjects who received Princess® FILLER Lidocaine AND the control Juvéderm® Ultra XC at the same visit as initial treatment; if subjects had received only one treatment (only Princess® FILLER Lidocaine or only Juvéderm® Ultra XC) during initial treatment they would have been excluded from the analysis set. Participants were analyzed as randomized. Only participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 249 | 249
Participants | 232 | 231

8. Secondary Outcome: Improvement Over Baseline Based on Subject Assessment at Week 24
Description: The percentage of subjects with an improvement over Baseline (subjects who have been rated as "very much improved" or "much improved" or "improved"), based on subject assessment at Week 24 after initial treatment and using the 5-point Global Aesthetic Improvement Scale (GAIS). GAIS grades are ranked as "very much improved", "much improved", "improved", "no change", and "worse".
Time Frame: Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Princess Filler Lidocaine | Comparator
Number analyzed (Participants) | 250 | 249
Participants | 229 | 228

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Groups:
- Blinded Period: Princess Filler Lidocaine: Treatment with Princess Filler Lidocaine: Injection into the nasolabial fold on either the left or the right side of the face.
- Blinded Period: Comparator: Treatment with Comparator: Injection into the nasolabial fold on either the right or the left side of the face.
- Open Label Extension Period: Princess Filler Lidocaine: Treatment with Princess Filler Lidocaine: Injection into the nasolabial fold on the left and the right side of the face.
Arm/Group | Blinded Period: Princess Filler Lidocaine | Blinded Period: Comparator | Open Label Extension Period: Princess Filler Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/270 | 0/48
Serious Adverse Events (participants affected / at risk) | 3/270 | 3/270 | 1/48
Other Adverse Events (participants affected / at risk) | 38/270 | 37/270 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Period: Princess Filler Lidocaine (N=270) | Blinded Period: Comparator (N=270) | Open Label Extension Period: Princess Filler Lidocaine (N=48)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Vascular compression (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Period: Princess Filler Lidocaine (N=270) | Blinded Period: Comparator (N=270) | Open Label Extension Period: Princess Filler Lidocaine (N=48)
COVID-19 (Infections and infestations) | 5 (5) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 12 (17) | 12 (17) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Swelling (General disorders) | 4 (4) | 2 (2) | 0 (0)
Discomfort (General disorders) | 3 (4) | 3 (3) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 0 (0)
Eyelid margin crusting (Eye disorders) | 6 (7) | 6 (7) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 4 (5) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 3 (4) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03990883/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT03990883/SAP_003.pdf